CLINICAL TRIAL: NCT02196753
Title: Positron Emission Tomography Combined With Computed Tomography (PET CT) in Suspected Cardiovascular Implantable Electronic Device Infection, a Pilot Study - PET Guidance I
Brief Title: PET CT in Suspected CIED Infection, a Pilot Study - PET Guidance I
Acronym: PET Guidance I
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Institute of Cardiology, Warsaw, Poland (Other)
Responsible Party: Sponsor
Other Study IDs: 2.32/V/2014
Record Dates: First submitted 2014-06-13; First posted 2014-07-22 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Complications; Infective Endocarditis; Implant Site Pocket Infection; Fever of Unknown Origin
Keywords: Positron emission tomography combined with computed tomography; PET CT; Cardiovascular Implantable Electronic Device; Infective endocarditis; Generator pocket infection; Fever of unknown origin
MeSH Terms: conditions — Endocarditis; Fever of Unknown Origin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- CIED related infection: All patients will undergo standard diagnostic process that will consist of: medical interview, physical examination, laboratory tests, blood cultures (3 sets, 1 hour apart, repeated after 24 hours and -if applicable - with fever peak above 38°C); imaging studies (echocardiography: transthoracic, and if there are no contraindications transesophageal, in case of negative or equivocal result repeated after 7-10 days, or in series if necessary, computed tomography scan for pulmonary embolism if indicated); if there are abnormalities in other systems, decisions concerning further diagnostics will be made by the physician in charge.
  Apart from standard diagnostic procedures patients will undergo whole body PET CT scan to localize infection or inflammation.
  Then the investigators team will make a decision concerning further treatment (antibiotics and complete device removal vs conservative treatment).
  Interventions: Other: PET CT
- Non-infective: Control group consisting of 20 pts with implanted CIEDs who underwent PET CT due to non infectious indications and have no data for infectious process in follow-up
  Interventions: Other: PET CT

INTERVENTIONS:
Other: PET CT — All patients are examined by a physicians before PET CT and if there are no contraindications they are given isotope intravenously. Then they stay in a warm waiting room. The dose of 18-FDG depends on patient's weight and varies from 270 to 420 MBq. Isotope uptake time is about 45-180 minutes. After that time the patient is asked to empty his or her bladder and go to the examination room. First CT scan lasting 2 min is performed followed by the PET scan lasting about 20 min. Usually area from mid tigh to eye level is scanned.
  In PET we use iterative reconstruction method (number of subsets 28, number of iterations 2), time of acquisition in one position of a table - 2 minutes. The following parameters will be analyzed: standardized uptake value (SUV) in the CIED area (pocket, leads), SUV of vascular background - pulmonary trunk, SUV of a liver, SUV max. in other potential changed areas, volume with increased SUV> 40% of the background.
  Other Names: Positron emission tomography - computed tomography

SUMMARY:
The aim of this single-center randomized controlled trial is to assess clinical usefulness of positron emission tomography combined with computed tomography (PET CT) in the diagnostic process of suspected cardiovascular implantable electronic device (CIED) infection (lead dependent infective endocarditis, generator pocket infection, fever of unknown origin).

DETAILED DESCRIPTION:
Cardiovascular implantable electronic device (CIED) infection is a complication of increasing incidence. The prevalence of CIED infection is estimated at 2%, with differences between authors ranging from 0.13% to 19.9%.

According to European Heart Rhythm Association survey conducted in high volume centers prevalence of CIED infections was below 2%. The majority of centers were able to isolate the infectious agent in ≤50% of blood cultures which underscore the difficulty in finding the agent of CIEDs infection in many cases.

Cardiovascular implantable device infections can be categorized into 3 groups: superficial skin infection, generator pocket infection and intravascular infection with intact generator pocket. Although local pocket infection is the most common clinical infection occurring early after implantation, positive blood cultures may be the only sign of late onset intravascular infection Mortality in cardiovascular implantable electronic device related infective endocarditis treated with antibiotics only reaches 66%, whereas with combined therapy (antibiotics and complete device removal) it is 3-fold lower.

Prolonged targeted antibiotic therapy (4 to 6 weeks) with complete device removal and revision of indications for re-implantation is recommended in most cases (class I with confirmed diagnosis and IIa with probable diagnosis).

In complicated and uncertain cases additional diagnostic tools are needed, especially if we take into account the load of the patient associated with device removal, prolonged hospitalization and re-implantation.

Apart from morbidity and mortality, infections are also associated with significant financial cost for patients and third-party payers. Polish data on this issue are not available yet but in US the estimated average cost of combined medical and surgical treatment of CIED-related infection ranges from USD 25,000 for permanent pacemakers to USD 50,000 for implantable cardioverter-defibrillators.

Positron emission tomography combined with computed tomography (PET CT) can play an important role in difficult cases of CIED-related infections but published studies focused on the outcomes and safety of this procedure only briefly considering the economical aspect of this diagnostic test.

Recent studies show that PET CT scan is effective and precise tool that can facilitate diagnostic process and decision making regarding therapy especially in difficult patients with CIED-related infections. PET CT scan can protect patients from unnecessary device removal or from too late removal. PET CT may also help in diagnosing other sources of infection, embolic complications, neoplasms, autoimmune diseases and connective tissue diseases.

However there are some issues concerning low sensitivity connected with elevated marker uptake in myocardium and in case of small vegetations, especially lead-related In most studies assessing PET CT in diagnostic process of CIED related infections standard oncologic protocols were used. Those protocols may not be optimal to assess FDG uptake by inflammatory cells.

The aim of this single-center randomized controlled trial is to assess clinical usefulness of positron emission tomography combined with computed tomography (PET CT) in the diagnostic process of suspected cardiovascular implantable electronic device (CIED) infection (lead dependent infective endocarditis, generator pocket infection, fever of unknown origin).

All patients participating in the study will undergo standard diagnostic process. Conventional/standard diagnostic and therapeutic process will consist of: medical interview, physical examination, laboratory tests, blood cultures (3 sets, 1 hour apart, repeated after 24 hours and -if applicable - with fever peak above 38°C); imaging studies (echocardiography: transthoracic, and if there are no contraindications transesophageal, in case of negative or equivocal result repeated after 7-10 days, or in series if necessary, computed tomography scan for pulmonary embolism if indicated); if there are abnormalities in other systems, decisions concerning further diagnostics will be made by the physician in charge.

Apart from standard diagnostic procedures patients will undergo whole body PET CT scan to localize infection or inflammation.

Then the investigators team will make a decision concerning further treatment (antibiotics and complete device removal vs conservative treatment).

ELIGIBILITY:
Inclusion Criteria:

* Age - 18 years and older.
* Written informed consent for participating in the study and written standard version of informed consent for PET CT scan.
* Suspected generator pocket infection
* Suspected cardiovascular implantable electronic device (CIED)-related infective endocarditis
* Fever of unknown origin in patient with CIED

Exclusion Criteria:

* Lack of written informed consent
* Pregnancy or breast feeding
* Inability to stay supine for the time of PET CT scan
* Unstable cardio-pulmonary state
* Glucose level above 200 mg/dl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study group - twenty pts with implanted CIEDs and suspected or diagnosed CIED-related infection or fever of unknown origin.
  Control group - twenty pts with implanted CIEDs who underwent PET CT due to non infectious indications and have no data for infectious process in follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2014-03; Primary Completion 2016-09 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants with established diagnosis | up to 6 months
  Standardization of PET CT in diagnostic process of local infections and lead dependent endocarditis in clinical practice. Sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV) of the diagnosis held by PET CT compared with final clinical diagnosis

SECONDARY OUTCOMES:
Number of participants with remote infective complications | up to 6 months
  Assessment of usefulness of PET CT for detection of remote infective complications (metastatic abscesses, infected pulmonary emboli)
Number of participants with particular localizations of infection | up to 6 months
  Incidence of particular localizations of infection
Number of participants with sustained therapuetic decision | up to 6 months
  Influence of PET CT on therapeutic decision: confirmation or change of decision based on PET CT (percentage)
Number of participants with complications of PET CT | up to 6 months
  Safety and complications of diagnostic process of CIED related infections with PET CT

CONTACTS AND LOCATIONS:
Overall Officials: Maciej Sterliński, MD, PhD, Principal Investigator — National Institute of Cardiology, Warsaw, Poland; Hanna Szwed, MD, PhD, Study Chair — National Institute of Cardiology, Warsaw, Poland
Locations (1):
- Institute of Cardiology, II Dept. of Coronary Heart Disease, Warsaw, Masovian Voivodeship, Poland

REFERENCES:
- [Background] Baddour LM, Epstein AE, Erickson CC, Knight BP, Levison ME, Lockhart PB, Masoudi FA, Okum EJ, Wilson WR, Beerman LB, Bolger AF, Estes NA 3rd, Gewitz M, Newburger JW, Schron EB, Taubert KA; American Heart Association Rheumatic Fever, Endocarditis, and Kawasaki Disease Committee; Council on Cardiovascular Disease in Young; Council on Cardiovascular Surgery and Anesthesia; Council on Cardiovascular Nursing; Council on Clinical Cardiology; Interdisciplinary Council on Quality of Care; American Heart Association. Update on cardiovascular implantable electronic device infections and their management: a scientific statement from the American Heart Association. Circulation. 2010 Jan 26;121(3):458-77. doi: 10.1161/CIRCULATIONAHA.109.192665. Epub 2010 Jan 4. PMID 20048212
- [Background] Klug D, Balde M, Pavin D, Hidden-Lucet F, Clementy J, Sadoul N, Rey JL, Lande G, Lazarus A, Victor J, Barnay C, Grandbastien B, Kacet S; PEOPLE Study Group. Risk factors related to infections of implanted pacemakers and cardioverter-defibrillators: results of a large prospective study. Circulation. 2007 Sep 18;116(12):1349-55. doi: 10.1161/CIRCULATIONAHA.106.678664. Epub 2007 Aug 27. PMID 17724263
- [Background] Greenspon AJ, Patel JD, Lau E, Ochoa JA, Frisch DR, Ho RT, Pavri BB, Kurtz SM. 16-year trends in the infection burden for pacemakers and implantable cardioverter-defibrillators in the United States 1993 to 2008. J Am Coll Cardiol. 2011 Aug 30;58(10):1001-6. doi: 10.1016/j.jacc.2011.04.033. PMID 21867833
- [Background] Cabell CH, Heidenreich PA, Chu VH, Moore CM, Stryjewski ME, Corey GR, Fowler VG Jr. Increasing rates of cardiac device infections among Medicare beneficiaries: 1990-1999. Am Heart J. 2004 Apr;147(4):582-6. doi: 10.1016/j.ahj.2003.06.005. PMID 15077071
- [Background] Bongiorni MG, Marinskis G, Lip GY, Svendsen JH, Dobreanu D, Blomstrom-Lundqvist C; Scientific Initiative Committee, European Heart Rhythm Association. How European centres diagnose, treat, and prevent CIED infections: results of an European Heart Rhythm Association survey. Europace. 2012 Nov;14(11):1666-9. doi: 10.1093/europace/eus350. PMID 23104858
- [Background] Dababneh AS, Sohail MR. Cardiovascular implantable electronic device infection: a stepwise approach to diagnosis and management. Cleve Clin J Med. 2011 Aug;78(8):529-37. doi: 10.3949/ccjm.78a.10169. PMID 21807925
- [Background] Habib G, Hoen B, Tornos P, Thuny F, Prendergast B, Vilacosta I, Moreillon P, de Jesus Antunes M, Thilen U, Lekakis J, Lengyel M, Muller L, Naber CK, Nihoyannopoulos P, Moritz A, Zamorano JL; ESC Committee for Practice Guidelines. Guidelines on the prevention, diagnosis, and treatment of infective endocarditis (new version 2009): the Task Force on the Prevention, Diagnosis, and Treatment of Infective Endocarditis of the European Society of Cardiology (ESC). Endorsed by the European Society of Clinical Microbiology and Infectious Diseases (ESCMID) and the International Society of Chemotherapy (ISC) for Infection and Cancer. Eur Heart J. 2009 Oct;30(19):2369-413. doi: 10.1093/eurheartj/ehp285. Epub 2009 Aug 27. No abstract available. PMID 19713420
- [Background] Darouiche RO. Treatment of infections associated with surgical implants. N Engl J Med. 2004 Apr 1;350(14):1422-9. doi: 10.1056/NEJMra035415. No abstract available. PMID 15070792
- [Background] Ferguson TB Jr, Ferguson CL, Crites K, Crimmins-Reda P. The additional hospital costs generated in the management of complications of pacemaker and defibrillator implantations. J Thorac Cardiovasc Surg. 1996 Apr;111(4):742-51;discussion 751-2. doi: 10.1016/s0022-5223(96)70334-3. PMID 8614134
- [Background] Farkowski MM, Milkowski M, Dziuk M, Pytkowski M, Marciniak M, Kraska A, Szwed H, Sterlinski M. Economical aspect of PET/CT-guided diagnosis of suspected infective endocarditis in a patient with implantable cardioverter-defibrillator. Heart Lung. 2014 Jul-Aug;43(4):341-3. doi: 10.1016/j.hrtlng.2014.04.002. Epub 2014 May 22. PMID 24856231
- [Background] Sarrazin JF, Philippon F, Tessier M, Guimond J, Molin F, Champagne J, Nault I, Blier L, Nadeau M, Charbonneau L, Trottier M, O'Hara G. Usefulness of fluorine-18 positron emission tomography/computed tomography for identification of cardiovascular implantable electronic device infections. J Am Coll Cardiol. 2012 May 1;59(18):1616-25. doi: 10.1016/j.jacc.2011.11.059. PMID 22538331
- [Background] Ploux S, Riviere A, Amraoui S, Whinnett Z, Barandon L, Lafitte S, Ritter P, Papaioannou G, Clementy J, Jais P, Bordenave L, Haissaguerre M, Bordachar P. Positron emission tomography in patients with suspected pacing system infections may play a critical role in difficult cases. Heart Rhythm. 2011 Sep;8(9):1478-81. doi: 10.1016/j.hrthm.2011.03.062. Epub 2011 Apr 2. PMID 21463705
- [Background] Bensimhon L, Lavergne T, Hugonnet F, Mainardi JL, Latremouille C, Maunoury C, Lepillier A, Le Heuzey JY, Faraggi M. Whole body [(18) F]fluorodeoxyglucose positron emission tomography imaging for the diagnosis of pacemaker or implantable cardioverter defibrillator infection: a preliminary prospective study. Clin Microbiol Infect. 2011 Jun;17(6):836-44. doi: 10.1111/j.1469-0691.2010.03312.x. Epub 2010 Jul 15. PMID 20636421
- [Background] Cautela J, Alessandrini S, Cammilleri S, Giorgi R, Richet H, Casalta JP, Habib G, Raoult D, Mundler O, Deharo JC. Diagnostic yield of FDG positron-emission tomography/computed tomography in patients with CEID infection: a pilot study. Europace. 2013 Feb;15(2):252-7. doi: 10.1093/europace/eus335. Epub 2012 Nov 12. PMID 23148119
- [Background] Leccisotti L, Perna F, Lago M, Leo M, Stefanelli A, Calcagni ML, Pelargonio G, Narducci ML, Bencardino G, Bellocci F, Giordano A. Cardiovascular implantable electronic device infection: delayed vs standard FDG PET-CT imaging. J Nucl Cardiol. 2014 Jun;21(3):622-32. doi: 10.1007/s12350-014-9896-2. Epub 2014 Apr 10. PMID 24715624
- [Background] Millar BC, Prendergast BD, Alavi A, Moore JE. 18FDG-positron emission tomography (PET) has a role to play in the diagnosis and therapy of infective endocarditis and cardiac device infection. Int J Cardiol. 2013 Sep 1;167(5):1724-36. doi: 10.1016/j.ijcard.2012.12.005. Epub 2013 Jan 11. PMID 23313465
- [Derived] Marciniak-Emmons MB, Swierzynska E, Mazurek A, Syska P, Farkowski MM, Firek B, Juszczyk U, Zakrzewska-Koperska J, Zajac D, Oreziak A, Maciag A, Kowalik I, Pytkowski M, Szwed H, Bilinska M, Szumowski L, Dziuk M, Sterlinski M. Computed tomography with positron emission tomography is more useful in local than systemic infectious process related to cardiac implanted electrotherapy device: a prospective controlled multicenter diagnostic intervention PET-Guidance Trial. Int J Cardiovasc Imaging. 2022 Dec;38(12):2753-2761. doi: 10.1007/s10554-022-02663-3. Epub 2022 Sep 7. PMID 36445676
- [Derived] Marciniak-Emmons MB, Sterlinski M, Syska P, Maciag A, Farkowski MM, Firek B, Dziuk M, Zajac D, Pytkowski M, Szwed H. New diagnostic pathways urgently needed. Protocol of PET Guidance I pilot study: positron emission tomography in suspected cardiac implantable electronic device-related infection. Kardiol Pol. 2016;74(1):47-52. doi: 10.5603/KP.a2015.0113. Epub 2015 Jun 23. PMID 26101020